CLINICAL TRIAL: NCT05259813
Title: An Open Label, Single-arm, Phase I Study of JWCAR029 in Subjects With Relapsed or Refractory Chronic Lymphocytic Leukemia or Small Lymphocytic Lymphoma
Brief Title: Phase I Study of JWCAR029 in Subjects With R/R CLL/SLL
Status: Withdrawn | Phase: Phase 1 | Type: Interventional
Why Stopped: Due to the COVID-19 pandemic，no subjects enrolled
Sponsor: Shanghai Ming Ju Biotechnology Co., Ltd. (Industry)
Collaborators: The First Affiliated Hospital with Nanjing Medical University (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: JWCAR029-007
Record Dates: First submitted 2022-02-08; First posted 2022-03-02 (Actual); Last update posted 2023-11-24 (Actual); Status verified 2023-11

CONDITIONS: Leukemia, Lymphocytic, Chronic, B-Cell
MeSH Terms: conditions — Leukemia, Lymphocytic, Chronic, B-Cell | interventions — relmacabtagene autoleucel

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- JWCAR029 Treatment (Experimental): Dose-finding for JWCAR029 monotherapy
  Interventions: Genetic: JWCAR029 (Relmacabtagene Autoleucel)

INTERVENTIONS:
Genetic: JWCAR029 (Relmacabtagene Autoleucel) — CD19-targeted Chimeric Antigen Receptor (CAR) T Cells

SUMMARY:
This is a Phase I, open-label, single-arm, single center study to assess the safety and efficacy of JWCAR029 in subjects With Relapsed or Refractory Chronic Lymphocytic Leukemia or Small Lymphocytic Lymphoma

DETAILED DESCRIPTION:
Upon the successful product generation of Relmacabtagene Autoleucel, subjects will enter the treatment phase of the study. Treatment will include lymphodepleting chemotherapy followed by Relmacabtagene Autoleucel administration. Subjects will then enter the post-treatment follow-up phase of the study and will be followed for approximately 24 months for safety, disease status, and survival. Long-term follow-up will continue under a separate long-term follow-up protocol, currently up to 15 years after the last Relmacabtagene Autoleucel administration.

ELIGIBILITY:
Inclusion Criteria:

* ≥ 18 years old and ≤ 75 years old;
* Sign on the informed consent;
* Diagnosis of:

  1. CLL with an indication for treatment based on iwCLL 2018 and measurable disease, or
  2. SLL (lymphadenopathy and/or splenomegaly and < 5×10^9 CD19+ CD5+ clonal B lymphocytes/L [< 5000/µL] in the peripheral blood at diagnosis with measurable disease that is biopsy-proven SLL);
* Relapsed/refractory patients, Subjects must have received and failed Bruton tyrosine kinase inhibitor (BTKi) treatment or have been deemed ineligible for BTKi therapy;
* Eastern Cooperative Oncology Group (ECOG) performance status of 0 or 1;
* Expected survival is greater than 12 weeks;
* Adequate organ function;
* Adequate vascular access for leukapheresis procedure;
* Women of childbearing potential must agree to use highly effective methods of contraception for 1 year after the last dose of JWCAR029; Males who have partners of childbearing potential must agree to use an effective barrier contraceptive method for 1 year after the last dose of JWCAR029.

Exclusion Criteria:

* Central nervous system (CNS) only involvement by malignancy or primary CNS lymphoma;
* History of another primary malignancy that has not been in remission for at least 2 years;
* Subjects has HBV, HCV, HIV or syphilis infection at the time of screening;
* Deep venous thrombosis (DVT)/Pulmonary embolism (PE), or DVT/PE requires anti-coagulation within 3 months prior to signing the ICF;
* Subjects with uncontrolled systemic fungal, bacterial, viral or other infection;
* Presence of acute or chronic graft-versus-host disease (GVHD);
* History of any serious cardiovascular disease or presence of clinically relevant CNS pathology;
* Pregnant or nursing women;
* Subjects using of any chemotherapy, corticosteriod, experiment agents, GVHD therapies, radiation or any other therapies for lymphoma must go through a specific wash-out period before leukapheresis;
* Received allo-hematopoietic stem cell transplantation therapy previously.
* Uncontrolled conditions or unwillingness or inability to follow the procedures required in the protocol;
* Received CAR T-cell or other genetically-modified T-cell therapy previously.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2022-02-28 (Estimated); Primary Completion 2023-01-31 (Estimated); Study Completion 2025-03-31 (Estimated)

PRIMARY OUTCOMES:
Treatment-related adverse events (AEs) | 2 years
  Type, Proportion, and Severity
Recommended dose of JWCAR029 | 28 days after JWCAR029 infusion
  Recommended dose of JWCAR029

SECONDARY OUTCOMES:
Best Objective response (BOR) rate | 3 months
  iwCLL2018
Best Complete response (CR) rate | 3 months
  iwCLL2018
Objective response rate (ORR) | 3 months
  iwCLL2018
Complete response rate (CRR) | 3 months
  iwCLL2018
MRD-negative response rate | 3 months
  Proportion of subjects who achieve MRD-negative OR and CR
Progression free survival (PFS) | 2 years
  iwCLL2018
Overall survival (OS) | 2 years
  iwCLL2018
Duration of response | 2 years
  iwCLL2018
Pharmacokinetics- Maximum concentration (Cmax) | 2 years
  Flow cytometry and qPCR
Pharmacokinetics- Time of the maximum concentration (Tmax) | 2 years
  Flow cytometry and qPCR
Pharmacokinetics- area under the curve | 2 years
  Flow cytometry and qPCR
Serum cytokines associated with CRS | 2 years
  IL-6, IL-8, TGF-β1, TNF-α, etc.

CONTACTS AND LOCATIONS:
Overall Officials: JianYong Li, Principal Investigator — The First Affiliated Hospital with Nanjing Medical University
Locations (1):
- Jiangsu Province Hospital, Nanjing, Jiangsu, China

IPD SHARING:
Plan to Share IPD: No